CLINICAL TRIAL: NCT07333274
Title: An Open-label, Prospective, Randomized, Phase III, International Multicenter Clinical Study to Compare Radiotherapy Plus Nimotuzumab Versus Radiotherapy Alone in Platinum-Ineligible Patients With Locoregionally Advanced Head and Neck Squamous Cell Carcinoma (LA-HNSCC)
Brief Title: Compare Radiotherapy Plus Nimotuzumab Versus Radiotherapy Alone in Platinum-ineligible Patients With Locoregionally Advanced Head and Neck Squamous Cell Carcinoma
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Shandong Cancer Hospital and Institute (Other)
Responsible Party: Principal Investigator, Man Hu, Shandong First Medical University Affiliated Cancer Hospital, Shandong Cancer Hospital and Institute
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IST-Nim-HNSCC-45
Record Dates: First submitted 2025-12-24; First posted 2026-01-12 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-12

CONDITIONS: Head & Neck Squamous Cell Carcinoma; Head & Neck Cancer
Keywords: Nimotuzumab; Radiotherapy; locoregionally advanced head and neck squamous cell carcinoma; LA-HNSCC
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Head and Neck Neoplasms | interventions — nimotuzumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Radiotherapy plus nimotuzumab (Experimental): radiotherapy plus nimotuzumab
  Interventions: Drug: Nimotuzumab; Radiation: intensity-modulated technique（IMRT）
- Radiotherapy alone in LA-HNSCC (Active Comparator)
  Interventions: Radiation: intensity-modulated technique（IMRT）

INTERVENTIONS:
Drug: Nimotuzumab — Treatment regimen： Nimotuzumab(Experimental Group): nimotuzumab injection 200 mg IV once weekly (QW) for 7 weeks (concurrent with radiotherapy).
  Other Names: Nimotuzumab injection
  Arms: Radiotherapy plus nimotuzumab
Radiation: intensity-modulated technique（IMRT） — Treatment regimen： Radiotherapy (both groups): intensity-modulated technique (photon IMRT or proton IMPT); total dose 70 Gy (2.0 Gy per fraction, 35 fractions), 5 fractions per week.
  Other Names: photon IMRT; proton IMPT; intensity-modulated technique

SUMMARY:
This is an open-label, prospective, randomized, Phase III, international multicenter clinical study to compare radiotherapy plus nimotuzumab versus radiotherapy alone in platinum-ineligible patients with locoregionally advanced head and neck squamous cell carcinoma (LA-HNSCC),

DETAILED DESCRIPTION:
This is an open-label, prospective, randomized, Phase III, international multicenter clinical study to compare radiotherapy plus nimotuzumab versus radiotherapy alone in platinum-ineligible patients with locoregionally advanced head and neck squamous cell carcinoma (LA-HNSCC), The study aims to evaluate the efficacy and safety of radiotherapy combined with nimotuzumab in platinum-ineligible patients with (LA-HNSCC).Around 70 study sites were involved in the trial.

ELIGIBILITY:
Inclusion Criteria:

* Eligible subjects must meet all of the following:

  * Age ≥18 years.
  * Histologically confirmed stage III-IVB (AJCC 8th edition) head and neck squamous cell carcinoma (including cancers of the oral cavity, oropharynx, hypopharynx, and larynx).
  * Unsuitable for surgical treatment (defined as: due to patient condition or tumor factors [T3-4 N0-3 M0, or T1-2 N2-3 M0] or medical reasons, surgery is not feasible; or an R0 resection is not achievable).
  * Suitable for definitive radiotherapy with curative intent.
  * At least one of the following reasons for being unsuitable for cisplatin-based chemotherapy:
* Age ≥65 years and, in the investigator's judgment, unable to tolerate chemotherapy;
* ECOG Performance Status >2 (if this criterion is met, the ECOG criterion listed below may be waived);
* Renal dysfunction: creatinine clearance (CrCl) <50 mL/min (Cockcroft-Gault) (if this criterion is met, the renal function criterion listed below may be waived);
* Severe tinnitus or hearing loss (requires a hearing aid or audiometry shows ≥25 dB loss at two consecutive frequencies);
* Peripheral neuropathy > Grade 1;
* Inability to receive intravenous hydration (e.g., due to cardiac dysfunction) or other comorbidities, per investigator's judgment.

  * Provide tumor tissue, whenever possible, for EGFR testing; for oropharyngeal cancer, provide tissue for HPV/p16 testing if feasible (no need to retest if previously tested).
  * ECOG Performance Status 0-1 (or Karnofsky Performance Status ≥80).
  * At least one measurable lesion per RECIST 1.1.
  * Expected survival ≥6 months.
  * Adequate hematologic function: WBC ≥4×10^9/L; absolute neutrophil count ≥1.5×10^9/L; platelets ≥100×10^9/L; hemoglobin ≥90 g/L.
  * Adequate renal function: serum creatinine ≤1.5×ULN or CrCl ≥60 mL/min (Cockcroft-Gault):
* Female CrCl = (140 - age) × weight (kg) × 0.85 / (72 × S_cr [mg/dL])
* Male CrCl = (140 - age) × weight (kg) × 1.00 / (72 × S_cr [mg/dL])

  * Adequate liver function: total bilirubin ≤1.5×ULN; AST ≤2.5×ULN; ALT ≤2.5×ULN.
  * Voluntary participation: signed written informed consent and ability to comply with visits and procedures.

Exclusion Criteria:

* Any of the following excludes enrollment:

  * Receipt of a PD-1 inhibitor, EGFR monoclonal antibody, EGFR-TKI, or anti-angiogenic agent within 4 weeks prior to enrollment.
  * Participation in another interventional clinical trial within 30 days prior to screening.
  * History of other malignancy (except cured basal cell carcinoma of the skin).
  * History of primary immunodeficiency.
  * Uncontrolled comorbid conditions (e.g., congestive heart failure, severe pulmonary disease, severe liver disease, psychiatric illness).
  * Known HIV infection, or active viral hepatitis or active tuberculosis.
  * Major surgery within 90 days before first study treatment, or planned surgery during the study.
  * Known allergy to nimotuzumab or its excipients.
  * Deemed unsuitable to participate by the investigator.
  * Unwilling or unable to sign informed consent.
  * Receipt of a live vaccine within 30 days before first dose.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 335 (Estimated)
Dates: Start 2026-01-05 (Estimated); Primary Completion 2028-01-05 (Estimated); Study Completion 2030-01-05 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) | 24 months after treatment initiation
  the proportion of patients in a clinical study who remain free of disease progression (including local recurrence, regional lymph node metastasis, distant metastasis, or second primary malignancy) and have not died from any cause within 2 years from the start of treatment (or randomization in randomized controlled trials).

SECONDARY OUTCOMES:
2-year locoregional control (LRC) rate. | 24 months after treatment initiation
  the proportion of patients in a clinical study who remain free of disease progression within 2 years from the start of treatment (or randomization in randomized controlled trials).
2-year distant metastasis rate. | 24 months after treatment initiation
  the prproportion of participants with distant metastatic progression within 24 months,
Overall Survival (OS) | 24 months after treatment initiation
  the prproportion of participants surviving at 2 years after enrolling,regardless of disease status.
Objective Response Rate (ORR; CR+PR by RECIST 1.1). | 24 months after treatment initiation
  the proportion of patients with measurable malignant tumors who achieve a complete response (CR) or partial response (PR)
Quality of Life (QoL) | 24 months after treatment initiation

CONTACTS AND LOCATIONS:
Overall Officials: Man Hu, Principal Investigator — Shandong First Medical University Affiliated Cancer Hospital
Locations (1):
- Shandong First Medical University Affiliated Cancer Hospital, Shandong, Province, China

IPD SHARING:
Plan to Share IPD: No